| Division | · | Worldwide Development |
|--------------------|---|-----------------------------------|
| Information Type : | | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for study 200196 A randomised double blind (sponsor unblinded), single and repeat ascending dose First Time in Human study in healthy subjects, cold urticaria and chronic spontaneous urticarial subjects to investigate safety, tolerability, pharmacodynamics and pharmacokinetics of GSK2646264 |
|---|---|---|
| <b>Compound Number</b> | : | GSK2646264 |
| <b>Effective Date</b> | : | 30-MAR-2015 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200196 [2013N167482 01].
- This RAP is intended to describe the safety, pharmacokinetics and pharmacodynamics analyses required for the study for Parts A, B and C.
- An informal interim review of the data following Part A, so as to provide project team and GSK stakeholders with key data to inform internal decision making, in order to start the Part B and C (cold urticaria and spontaneous urticaria subjects) of this study will be performed.
- This RAP will be provided to the study team members to convey the content of the [Reference as Required: Statistical Analysis Complete (SAC)] deliverable.

#### Author's Name and Functional Area:

| PPD | 30-MAR-2015 |
|-------------------------------------------------|-------------|
| Principal Biostatistician (PAREXEL Early Phase) | 30-MAK-2013 |

#### Approved by:

| PPD | | 30-MAR-2015 |
|--------------|------------------|-------------|
| Manager, Cli | nical Statistics | 30-MAK-2013 |

Copyright 2015 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS | S PLAN SYNPOSIS | 5 |
| 2. | SUMM<br>2.1. | | | TOCOL INFORMATIONtocol Defined Statistical Analysis Plan | |
| | 2.2.<br>2.3. | Study O | bjective(s) | and Endpoint(s) | <mark>7</mark> |
| | 2.4. | | | ses | |
| 3. | 3.1. | Interim A | Analysis (In | formal Data review) | 10 |
| | 3.2. | Final An | alyses | | 11 |
| 4. | ANAL`<br>4.1. | | | S | |
| 5. | | | | DATA ANALYSES AND DATA HANDLING | 13 |
| 6. | | | | ALYSES | |
| | 6.1. | Overvie | w of Planne | ed Analyses | 13 |
| 7. | PRIMA<br>7.1. | | | ANALYSES | |
| | , | 7.1.1. | Overview | of Planned Analyses | 14 |
| | | | 7.1.1.1. | Dose Escalations | 15 |
| 8. | | | | AL ANALYSES | |
| | 8.1. | 8.1.1. | | nalysescentration Measures | |
| | | 8.1.1.<br>8.1.2. | | okinetic Parameters | |
| | | 0.1.2. | 8.1.2.1. | Deriving Pharmacokinetic Parameters | |
| | | | 8.1.2.2. | Statistical Analysis of Pharmacokinetic | |
| | | | | Parameters | |
| 9. | EXPL( | | | TCAL ANALYSIS | |
| | 9.1. | | | and Biomarker Analyses | |
| | | 9.1.1. | | of Planned Pharmacodynamic Analyses | |
| | | 9.1.2. | | Pharmacodynamic Statistical Analyses | 19 |
| | | | 9.1.2.1. | Part C: Chronic Spontaneous Urticaria Subjects | 19 |
| | | | 9.1.2.2. | The Angioedema Activity Score (AAS) | 19 |
| | | | 9.1.2.3. | Relationships between Basophil Histamine | |
| | | | 5 | Release (BHR) Test and Weal Characteristics | |
| | | 9.1.3. | | Health Outcome Statistical Analyses | 21 |
| | | | 9.1.3.1. | Health Outcomes Analyses/ Dermatology Life | 24 |
| | | 9.1.4. | Overview | Quality Indexof Planned Biomarker Analyses | 21 |
| | 9.2. | | | and Biomarker Analyses | |
| | 0.2. | . Hallila | | and Bromainor Analyses | |


| 2 | $\sim$ | ١4 | $\sim$ | _ |
|---|--------|-----|--------|---|
| | ດເ | ) I | м | n |

| 0. | REFE | RENCES | | .23 |
|---|---|---|---|---|
| 11. | APPEN | NDICES | | .24 |
| | 11.1. | <b>Appendix</b> | c 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | . 25 |
| | | | predefined Populations | .25 |
| | 11.2. | Appendix | c 2: Time & Events | . 26 |
| | | 11.2.1. | Protocol Defined Time & Events | |
| | | | 11.2.1.1. Part A, Dose Group 1 (Healthy Volunteers) | .26 |
| | | | 11.2.1.2. Part A: Healthy Volunteer Time and Event | |
| | | | Table Dose group 2 | |
| | | | 11.2.1.3. Part B (Cold Urticaria Subjects) | |
| | | | 11.2.1.4. Part C (Chronic Spontaneous Urticaria Cohort) | .32 |
| | 11.3. | | 3: Data Display Standards & Handling Conventions | |
| | | 11.3.2. | Baseline Definition & Derivations | |
| | | | 11.3.2.1. Baseline Definitions | .36 |
| | | | 11.3.2.2. Derivations and Handling of Missing Baseline | <b>~</b> |
| | | 44.0.0 | Data | |
| | 44.4 | 11.3.3. | Reporting Process & Standards | .37 |
| | 11.4. | | 4: Derived and Transformed Data | |
| | 44.5 | | | |
| | 11.5. | | 5: Premature Withdrawals & Handling of Missing Data | |
| | | 11.5.2. | Handling of Missing Data | .43 |
| | | | 11.5.2.1. Handling of Missing Dates | |
| | 44.0 | ۸ا! | 11.5.2.2. Handling of Partial Dates | |
| | 11.6. | | (6: Values of Potential Clinical Importance | |
| | | | , | |
| | 44 7 | | Vital Signs | |
| | 11.7. | | 7: Examination of Covariates, Subgroups & Other Strata | |
| | 44.0 | | Handling of Covariates, Subgroups & Other Strata | .48 |
| | 11.8. | | x 8: Model Checking and Diagnostics for Statistical | 40 |
| | | | Statistical Anglysis Assumptions | |
| | 11.0 | | , i | |
| | 11.9. | | ( 9: Abbreviations & Trade Marks | |
| | | - | Trademarks | |
| | 11 10 | | ( 10: List of Data Displays | |
| | 11.10. | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverable [Priority] | |
| | | | Study Population Tables | |
| | | | Efficacy Tables | |
| | | | Safety Tables | |
| | | | Safety Figures | |
| | | 11.1U.Ö. | Pharmacokinetic Tables | . ၁9 |


| 11.10.9. Pharmacokinetic Figures | 60 |
|-----------------------------------------------------------|------------------|
| 11.10.10.Pharmacodynamic and Biomarker Tables | |
| 11.10.11.Pharmacodynamic Figures | |
| 11.10.12.ICH Listings | |
| 11.10.13. Non-ICH Listings | <mark>7</mark> 4 |
| 11.11. Appendix 11: Example Mock Shells for Data Displays | |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this RAP is to describe: |
| | An informal interim analysis, so as to provide project team and GSK stakeholders with key data to inform internal decision making, in order to start the Part B and C (cold urticaria and spontaneous urticaria subjects) of this study. |
| | This RAP will be provided to the study team members to convey the content of the [Reference as Required: Statistical Analysis Complete (SAC)] deliverable. |
| Protocol | This RAP is based on the protocol amendment 2 [(Dated: 10/DEC/2014) of study GSK2646264 (GSK Document Number: 2013N167482_01] and eCRF Version (Version 1, 09OCT2014). |
| Primary<br>Objective | The primary objective is to investigate the safety and tolerability of topically applied GSK2646264 cream and its placebo in healthy subjects, subjects with cold urticaria (CU) and subjects with chronic spontaneous urticaria (CsU) |
| Primary<br>Endpoint | Safety and Tolerability (Number, severity and frequency of AEs and serious AEs (local and systemic), heart rate, blood pressure, 12- lead ECG, clinical laboratory safety tests, assessment of the local tolerability of the study medication |
| Study<br>Design | Randomised, double blind (sponsor unblinded), bilateral, single and repeat ascending dose First Time in Human study in healthy subjects, cold urticaria and chronic spontaneous urticaria subjects. |
| | <ul> <li>Approximately 18 randomised evaluable subjects in Part A, and approximately<br/>12 randomised evaluable subjects in part B and C of study.</li> </ul> |
| Planned<br>Analyses | Safety and Tolerability, PK, PD (Allergen challenge, UAS7, AAS), Health Outcome (DLQI) |
| Analysis | Primary: Safety population, |
| Populations | Other: PK, PD, Per-Protocol populations |
| Hypothesis | There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | Safety data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| Secondary<br>Analyses | <ul> <li>Individual GSK2646264 plasma concentration-time profiles and median/mean<br/>(±SD) profiles will be plotted and listed. Plasma concentration time data for<br/>GSK2646264 will be analyzed by non-compartmental methods using WinNonlin<br/>and derived PK parameters (AUC, C<sub>max</sub>, T<sub>max</sub>, t<sub>1/2</sub>) summarized, listed and<br/>plotted. No formal statistical analyses will be conducted.</li> </ul> |
| Exploratory<br>Analyses | All PD endpoints will be summarized, listed and graphically presented. Where |


| Key Elements of the RAP |
|---|
| applicable, Paired t-Tests and/or ANCOVA model will be performed. Point estimates, and 95% confidence interval will be provided. |
| <u> </u> |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The following changes or deviations to the originally planned statistical analysis specified in the protocol [(Dated: 10/DEC/2014)].

- Study endpoints were modified for Part A of the study as some of the data points mentioned in original planned protocol analyses were not feasible to obtain via method and equipment used in the study.
- After Dose escalation meeting (at the end of dose group 1), dosing of dose group 2 in Part A study was modified. In a new design, subjects will be dosed up to 4 days only and up to a maximum BSA level of 10% in order to further understand the elimination phase of the systemic drug concentration. Therefore, all analyses will be carried out using new dosing plan.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Part A, B and C | Part A, B and C |
| To investigate the safety and tolerability of topically applied GSK2646264 cream and its placebo in healthy¹ subjects, subjects with cold urticaria (CU¹) and subjects with chronic spontaneous urticaria (CsU). | <ul> <li>Number, severity and frequency of AEs and serious AEs (local and systemic)</li> <li>Heart rate</li> <li>Blood pressure</li> <li>12- lead ECG</li> <li>Clinical laboratory safety tests</li> <li>Assessment of the local tolerability of the study medication</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| Part A, B and C | Part A, B and C |
| To evaluate the plasma<br>concentrations of GSK2646264 in<br>Healthy, CU and CsU subjects | <ul> <li>Plasma concentrations of GSK2646264 and<br/>pharmacokinetic parameters, including AUC, C<sub>max</sub>, T<sub>max</sub>,<br/>t<sub>1/2</sub>, if data allows</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| Part A: Healthy Subjects | Part A: Healthy Subjects |
| <ul> <li>Assess the pharmacodynamic effect of GSK2646264 on weal and flare sizes and erythema, in healthy subjects after allergen challenge (Skin Prick test, positive control (histamine) and negative control (Saline)).</li> <li>Duration of response in healthy subjects</li> </ul> | <ul> <li>Percent inhibition on days 1, 3, 4 and 6<sup>6</sup> for the longest weal diameter (measured by ruler).</li> <li>Percent inhibition on days 1, 3, 4 and 6<sup>6</sup> for perpendicular weal length (measured by ruler).</li> <li>Percent inhibition on days 1, 3, 4 and 6<sup>6</sup> for weal area (calculated<sup>5</sup>).</li> <li>Percent inhibition on days 1, 3, 4 and 6<sup>6</sup> for Weal volume (measured by quantitative volumetric morphometry<sup>2</sup>)</li> <li>Percent inhibition on days 1, 3, 4 and 6<sup>6</sup> for Flare erythema (measured by Mexameter<sup>3</sup>).</li> <li>Percent of inhibition at 48 hours post final dose, will be derived for the endpoints above</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Part B: Cold Urticaria Subjects | Part B: Cold Urticaria Subjects |
| To assess the pharmacodynamic effect of GSK2646264 on weal and flare sizes and erythema, in cold urticaria subjects after allergen challenge (Skin Prick test, positive control (histamine) and negative control (Saline)). | <ul> <li>Percent inhibition on days 1, and 3 for the longest weal diameter (measured by ruler).</li> <li>Percent inhibition on days 1, and 3 for perpendicular weal length (measured by ruler).</li> <li>Percent inhibition on days 1, and 3 for weal area (calculated).</li> <li>Percent inhibition on days 1, and 3 for Weal volume (measured by quantitative volumetric morphometry¹)</li> <li>Percent inhibition on days 1, and 3 for Flare erythema (measured by Mexameter²).</li> </ul> |
| To assess the effect of GSK2646264<br>on Cold Temperature Test values Part C: Chronic Spontaneous Urticaria | Change in Cold Temperature Test <sup>4</sup> values at day 1 and day 3 Part C: Chronic Spontaneous Urticaria Subjects |
| Subjects | |
| To assess the effect of GSK2646264<br>on weal characterisation in CsU<br>subjects within treated area only | <ul> <li>Urticaria Activity Score, a composite score using key<br/>urticaria symptoms (number of weals, Itch/Pruritus), to<br/>derive change from baseline on Day 1 through to Day 7</li> </ul> |
| <ul> <li>To assess the Quality of Life in CsU<br/>subjects.</li> </ul> | <ul> <li>Change from baseline in total Dermatology Life Quality<br/>Index (DLQI) score</li> </ul> |
| <ul> <li>To assess the disease activity in CsU subjects.</li> </ul> | Change from baseline in Angioedema Activity Score (AAS) |
| To investigate the relationships<br>between (basophil histamine release)<br>BHR test and weal characteristics | Relationship of positive BHR test with reduction in number or size of weals ects should be screened for reactivity to one of the allergens used in |

<sup>1</sup> All Healthy subjects and the Cold Urticaria subjects should be screened for reactivity to one of the allergens used in skin prick test. (grass pollen, Dermatophagoides pteronyssinus, birch pollen and cat dander)

<sup>2</sup> Measured using digital camera using PRIMOS 5.075D instrument software produced by GMF

<sup>3</sup> Measures erythema and melanin index values using narrow band spectrophotometry

<sup>4</sup> TEMPTest 4.0

<sup>5</sup> Calculated as ellipse or oval area

#### 2.3. Study Design



| Overview of Stu | dy Design and Key Features |
|---|---|
| | <ul> <li>Part A dosing group 2</li> <li>Part B</li> <li>Part C</li> <li>Each sentinel subject will be dosed at least 1 day before any other subjects of their dosing group or cohort.</li> <li>Subjects will be assigned to treatment in accordance with the randomization schedule using IVRS system. Randomisation will occur within each cohort of study. Each subject will be randomised to receive bilateral treatment of GSK2646264 or placebo. Randomisation will assign active and placebo to specified areas on left or right side of the body. The left or right side assignment of treatment always refers to the subject's left or right.</li> </ul> |
| Interim<br>Analysis<br>Informal data<br>review | <ul> <li>No formal interim analyses are planned.</li> <li>An informal summary of the safety, tolerability, PK and PD data from Part-A will be performed once all subjects are recruited and completed all visits.</li> </ul> |

# 2.4. Statistical Hypotheses

The primary focus of the statistical analysis is to describe safety and characterize the preliminary pharmacokinetics of GSK2646264 through estimates of parameters and their variability. Thus, an estimation approach will be taken and 95% confidence intervals will be constructed to provide a plausible range of values, where appropriate, with no formal hypothesis testing. Sample size estimations and results of succeeding sensitivity analyses are given in 9.2 of the protocol.

#### 3. PLANNED ANALYSES

# 3.1. Interim Analysis (Informal Data review)

No formal interim analyses are planned.

| Analysis | Definition / Criteria Analyses Evaluated |
|---|---|
| During the study | There will be ongoing data reviews conducted by the study team of the unblinded safety and pharmacodynamic data, and any available pharmacokinetic data throughout the trial progression. |
| Dose Escalation | Dose escalation meetings will be performed as stated in the protocol. At the end of dosing group 1 in Part A, the decision to proceed to the next higher strength and dose for dosing group 2 will be made by the SMC based on a safety report from the PI or designee, on the clinical safety, tolerability, up to and including the follow up visit, and pharmacokinetic exposure up to 24 hours after the last dose, in at least 6 subjects at the highest dose level. The GSK review team will be unblinded to the randomisation code and will usually include the GSK pharmacokineticist, GSK statistician, GSK data management, GSK medical monitor, GSK study team leader, GSK Global Clinical Safety and |

| Analysis | Definition / Criteria Analyses Evaluated |
|---|---|
| | Pharmacovigilance and GSK Clinical Matrix Team leader. |
| Part A<br>Completion | A summary of the safety, tolerability, PK and PD data from Part-A will be performed once all subjects are recruited and completed all visits. This summary will include PK and PD data from Part-A of study cohort. All safety data including adverse events, tolerability, laboratory tests, ECGs and vital signs will be reviewed. The decision to proceed to Part B and C will be made by the investigator and the GSK SMC review team based on assessment of safety and pharmacokinetic data of the studied doses. |

The Investigator or designee, study coordinators and any other unit staff who have been involved in assessing subjects will remain blinded during the study; however, they will attend the start of each review meeting to update the GSK team on safety and tolerability summary from each cohort; these team members will not be part of the unblinded dose escalation discussions. The investigator and/or designee should send the relevant data to the GSK review team prior to the meeting of the Safety Monitoring Committee (SMC). The study monitor will remain blinded.

The Safety Monitoring Committee (SMC) will consist of the GSK review team and the Investigator and/or designee. (See Section 5.5. of the protocol for further information)

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed (including for those subjects who withdrew or were withdrawn) the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database released.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to procedure.
- 5. Database freeze has been declared by Data Management

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety Population | Comprise of subjects who receive at least one dose of study medication. | Study Population Safety |
| | | • |
| Pharmacokinetic<br>(PK) Population | Comprise of all randomised subjects of the Safety Population for whom a pharmacokinetic sample was obtained and analysed. | PK-Analyses |
| Pharmacodynamic (PD) Population | Comprise of all randomised subjects of the Safety Population for whom a pharmacodynamic measurement sample was obtained and analysed. | PD -Analyses |
| | measurement sample was obtained and analysed. Analysis will be based on the actual treatment the subject received for the assigned area | |
| Per-Protocol | Comprise of all PD population subjects who | As required for PD- |
| Population | <ul> <li>receive at least one dose of study treatment and who comply with the protocol.</li> <li>Protocol deviations that would exclude subjects from the PP population are defined in Appendix 1 (Protocol Deviation Management Plan) for Definition Per-Protocol Population).</li> </ul> | Analyses |

#### NOTES:

 Please refer to Appendix 10: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population)].
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviations Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised in the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

 A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned examination of covariates and subgroups.
- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 11.4 | Appendix 4: Derived and Transformed Data |
| 11.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 11.6 | Appendix 6: Values of Potential Clinical Importance |
| 11.7 | Appendix 7: Examination of Covariates, Subgroups & Other Strata |
| 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |
| 11.9 | Appendix 9: Abbreviations & Trade Marks |
| 11.10 | Appendix 10: List of Data Displays |
| 11.11 | Appendix 11: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses for Part A, B and C of study

| [Endpoint / Parameter / Display Type] | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomisation | | | |
| Randomisation | | | Y |
| Disposition | | | |
| Subject Disposition | Y | | |
| Investigational Product Status | Y | | |
| Reasons for screen failure | | | Y |
| Reasons for withdrawals | | | Y |
| Important Protocol Deviations | Y | | Y |
| Deviation leading to exclusion from PP population | | | Y |
| Inclusion and exclusion criteria deviation | | | Υ |
| Study Population | Y | | |
| Demographics | | | |
| Demographic Characteristics | Y | | Υ |
| Race and Racial Combinations | Y | | Y |
| Medical History | | | |
| Medical History | Y | | Y |
| Concomitant Medication | | | |
| Concomitant Medication | Y | | Υ |

### 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Safety Analyses

#### 7.1.1. Overview of Planned Analyses

The safety analyses will be based on the 'Safety' population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Safety Analyses for Part A, B and C of study

| Endpoint / Parameter/ | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type | Sum | mary | Indiv | ridual | Sum | mary | Individual | |
| | Т | F | F | L | Т | F | F | L |
| Drug Exposure | | | | | | | | |
| Exposure to Study | Υ | | | Υ | | | | |
| Drug | | | | | | | | |
| Adverse Events | | | | | | | | |
| Summary of All | Υ | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| Drug-Related Adverse | Y | | | | | | | |
| Events | | | | | | | | |

<sup>•</sup> Y = Yes display generated.

| Endpoint / Parameter/ | | Abso | olute | | | Change fro | m Baselin | е |
|---|---|---|---|---|---|---|---|---|
| Display Type | Sum | mary | Indiv | idual | Sum | mary | Indiv | idual |
| | T | F | F | L | Т | F | F | L |
| Summary of All | Υ | | | | | | | |
| Localised Adverse | | | | | | | | |
| Events | | | | | | | | |
| Serious Adverse | Υ | | | Υ | | | | |
| Events | | | | | | | | |
| AEs Leading to | Υ | | | Υ | | | | |
| Discontinuation | | | | | | | | |
| AE by Maximum | Υ | | | | | | | |
| Intensity | | | | | | | | |
| Clinical Laboratory Ass | sessments | , | | | | | | |
| Clinical Chemistry | Υ | | | Υ | Υ | | | Υ |
| Haematology | Υ | | | Υ | Υ | | | Υ |
| Urinalysis | Υ | | | <b>Y</b> 1 | Υ | | | |
| Electrocardiogram (EC | <b>G</b> ) | | | • | | | | |
| ECG Findings | Υ | | | Υ | Υ | | | Υ |
| ECG Values | Υ | | | Υ | Υ | | | Υ |
| Vital Signs | | | | | | | | |
| Vital Signs | Υ | | | Υ | Υ | | | Υ |
| Tolerability assessmen | t | | | | | | | |
| Tolerability scores | Υ | | | Υ | Υ | | | Υ |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Tolerability analyses will be produced for Part A and B only.
  - 1 Urinalysis will only list abnormal assessments

#### 7.1.1.1. Dose Escalations

The principal investigator and study monitor will provide a report of findings during the last treatment for progressing to the next cohort, as defined in the protocol, but remain blinded. As required, ongoing data reviews will be conducted by the unblinded GSK study team throughout the trial progression.

#### 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic population, unless otherwise specified.

Table 4 provides an overview of the planned analyses, with full details being presented in Appendix 10: List of Data Displays

Table 4 Overview of Planned Pharmacokinetic Analyses for Part A, B and C of study

| Endpoint / Parameter/ | | | Untr | ransfo | rmed | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis | | Summary Inc | | Indiv | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Pharmacokinetics | | | | | | | | | | | | | | |
| PK concentrations | | | | Υ | Υ | Υ | Υ | | | | | | Υ | |
| PK parameters | | | | Υ | | | Υ | | | | Υ | | | |

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Process & Standards).

#### 8.1.2. Pharmacokinetic Parameters

#### 8.1.2.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix : Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WNL v6.3.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in **** Table 5 will be determined from the plasma concentration-time data, as data permits.

Table 5 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-24) | Area under the concentration-time curve from time zero to 24 hours after dosing |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| %AUCex | The percentage of AUC (0-∞) obtained by extrapolation (%AUCex) will be calculated as: [AUC(0-inf) – AUC(0-t)] / AUC(0-inf) x 100 |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: t½ = ln2 / lambda_z |

- Additional parameters may be included as required.
- Lambda z is the terminal phase rate constant.

#### 8.1.2.2. Statistical Analysis of Pharmacokinetic Parameters

All the derived parameters described above will be listed. The first point, last point and number of points used in the determination of  $\lambda_z$  will be included on the listing of the derived parameters. For each of the PK parameters, except  $t_{max}$  and %AUC<sub>wextrap</sub>, the following summary statistics will be calculated for each active treatment group: median, maximum, minimum, arithmetic mean, standard deviation, coefficient of variation, geometric mean, 95% confidence interval for the geometric mean and standard deviation of logarithmically transformed data. For  $t_{max}$  and %AUC<sub>wextrap</sub>, median, maximum, minimum, arithmetic mean and standard deviation will be calculated. All statistical analysis results of these PK parameters will be presented in relation to the actual dose given (i.e. the BSA covered)

### 9. EXPLORATORY STATISTICAL ANALYSIS

#### 9.1. Pharmacodynamic and Biomarker Analyses

#### 9.1.1. Overview of Planned Pharmacodynamic Analyses

The pharmacodynamic analyses will be based on the 'Pharmacodynamic' and Perprotocol populations, unless otherwise specified. All summaries will be presented by treatment group and/or include total column. Figures comparing the different treatments will be displayed overlayed where possible.

• If endpoints are listed, then all data will be listed.

Table 6 provides an overview of the planned pharmacodynamic analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 6 Overview of Planned Pharmacodynamic Analyses for Part A

| [Endpoint / | | Untransformed | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | | P | bsolu | bsolute | | | | Percent of Inhibition | | | | | |
| Type] | Stat | s Ana | lysis | Sum | mary | Indiv | ividual Stats A | | | lysis | Sum | nmary Indiv | | ridual |
| | T | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| Allergen Challenge - Pa | Allergen Challenge - Part A : Healthy Subjects | | | | | | | | | | | | | |
| Weal area (mm²) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Weal volume (mm <sup>3</sup> ) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Longest Weal diameter (mm) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Weal perpendicular length (Height) (mm) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Flare erythema ((mm²) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data. Summary will be presented by dose strength, BSA and day (if applicable)
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Weal area derived from weal longest diameter and perpendicular length; assuming elliptic shape.

Table 7 Overview of Planned Pharmacodynamic Analyses for Part B

| [Endpoint / | Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | | Δ | bsolu | ite | | | Percent of Inhibition/Change 1 | | | | | | |
| Type] | Stat | s Ana | lysis | Sum | mary | Indiv | Individual | | Stats Analysis | | | Summary | | Individual |
| | Т | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| Allergen Challenge - Part B: Cold Urticaria Subjects | | | | | | | | | | | | | | |
| Weal area (mm <sup>2</sup> ) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Weal volume (mm <sup>3</sup> ) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Weal longest diameter (mm) | | | | Υ | Υ | | Y | | | | Υ | Υ | Υ | Υ |
| Weal perpendicular length (Height) (mm) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Flare erythema ((mm²) | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |
| Cold Temperature Test | | | | Υ | Υ | | Υ | | | | Υ | Υ | Υ | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Summary will be presented by dose strength, BSA and day (if applicable)
- 1. Change will be produced for Cold Tem Test endpoint

Table 8 Overview of Planned Pharmacodynamic Analyses for Part C

| [Endpoint / | | | | | | U | ntrans | sform | ed | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | | A | bsolu | ite | | | Change from Baseline | | | | | | |
| Type] | Stat | s Ana | lysis | Sum | mary | Indiv | Individual | | Stats Analysis | | | mary | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | Г |
| Pharmacodynamic - Part C: Chronic Spontaneous Urticaria Subjects | | | | | | | | | | | | | | |
| UAS7 score | | | | Υ | | | Υ | Υ | | | Υ | Υ | | Υ |
| Angioedema Activity | | | | V | | | V | V | | | V | V | | \<br>\ |
| Score (AAS | | | | T | | | I | ľ | | | T | ĭ | | ĭ |
| UAS7 components | | | | | | | | | | | | | | |
| (Number of weals, | | | | Υ | | | Υ | Υ | | | Υ | Υ | | Υ |
| Extent of Itch) | | | | | | | | | | | | | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Summary will be presented by dose strength, BSA and day (if applicable)

### 9.1.2. Planned Pharmacodynamic Statistical Analyses

#### 9.1.2.1. Part C: Chronic Spontaneous Urticaria Subjects

## **Planned Statistical Analyses**

#### Endpoint(s)

• Change from baseline in composite total UAS7 score and components

#### Model Specification

- Endpoint will be analysed using paired t test and ANCOVA to compare the treatment groups.
- ANCOVA model will be fitted as: Post-Pre dose as response and pre dose as covariate.

#### **Model Checking**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Estimated treatment difference and 95% confidence intervals will be presented.

#### **Analysis of UAS7 Components**

- Analysis of UAS7 components will be performed similar to total UAS7 composite score
- Summary Statistics for each component of UAS7 questionnaire will be provided by visit.

#### Note:

- Composite score UAS7 will be derived using key urticaria symptoms (number of weal, Itch/Pruritus). The UAS7 score will be calculated using the summation of the 7 consecutive days sum.
- Other questions collected as part of UAS7 questionnaire will be listed.

#### 9.1.2.2. The Angioedema Activity Score (AAS)

#### **Planned Statistical Analyses**

#### **Planned Statistical Analyses**

#### Endpoint(s)

• Change from baseline in total and individual item score

#### **Model Specification**

- Endpoint will be analyzed using paired t test and ANCOVA to compare the treatment groups.
- ANCOVA model will be fitted as: Post-Pre dose as response and pre dose as covariate.

#### **Model Checking**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• Estimated treatment difference and 95% confidence intervals will be presented.

#### **Analysis of AAS Components**

Summary Statistics for each component AAS questionnaire will be provided by visit.

#### Note:

Details of the Angioedema Activity Score (AAS) questionnaire are provided in Appendix 7
of the protocol. Each AAS item will be scored between 0 to 3 and daily total score AAS
score will range between 0 and 15. The daily AAS score will be summed up to compute 7day total scores

# 9.1.2.3. Relationships between Basophil Histamine Release (BHR) Test and Weal Characteristics

#### **Planned Statistical Analyses**

#### Endpoint(s)

Positive BHR Test

#### **Model Specification**

• Endpoint will be analyzed using logistic regression with weal characteristics (i.e. weal length) as covariate to establish the relationship between BHR test and weal characteristics.

#### **Model Checking**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Odds Ratio and 95% Confidence intervals

## 9.1.3. Planned Health Outcome Statistical Analyses

#### Table 9 Overview of Planned Health Outcome Analyses for Part C

| [Endpoint / | | Untransformed | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | | A | Absolu | te | | | Change from Baseline | | | | | | |
| Type] | Stat | Stats Analysis Summary Individual | | | | | | | s Ana | lysis | Sum | mary | Individual | |
| | Τ | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Health Outcome - Part | C: Ch | ronic | Spor | taneo | us Ur | ticaria | Subje | ects | | | | | | |
| Dermatology Life<br>Quality Index (DLQI) | | | | Υ | Y | | Y | Υ | | | Υ | Υ | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Summary will be presented by dose strength, BSA and day (if applicable)

#### 9.1.3.1. Health Outcomes Analyses/ Dermatology Life Quality Index

| Planned Statistical Analyses | |
|---|---|
| Endpoint(s) | |
| Change from baseline in total and individual domain scores | |
| Model Specification | |
| <ul> <li>Endpoint will be analyzed using paired t te</li> </ul> | Endpoint will be analyzed using paired t test to compare the improvement in quality of life |
| Model Checking | |
| <ul> <li>Refer to Appendix 8: Model Checking and</li> </ul> | Diagnostics for Statistical Analyses. |
| Model Results Presentation | |
| <ul> <li>Estimated treatment difference and 95% of the state of th</li></ul> | confidence intervals will be presented. |
| Very much | scored 3 |
| A lot | scored 2 |
| A little | scored 1 |
| Not at all | scored 0 |
| Not relevant | scored 0 |
| Question unanswered scored 0 | |
| Question 7: "prevented work or studying" scored 3 | |
| <ul> <li>The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.</li> <li>The six subscores will be derived as follows:</li> </ul> | |

| Planned Statistical Analyses | | |
|------------------------------|-------------------|-----------------|
| Symptoms and feelings | Questions 1 and 2 | Score maximum 6 |
| Daily activities | Questions 3 and 4 | Score maximum 6 |
| Leisure | Questions 5 and 6 | Score maximum 6 |
| Work and School | Question 7 | Score maximum 3 |
| Personal relationships | Questions 8 and 9 | Score maximum 6 |
| Treatment | Question 10 | Score maximum 3 |

#### 9.1.4. Overview of Planned Biomarker Analyses

The biomarker analyses will be based on the 'Pharmacodynamic' population, unless otherwise specified.

Table 10 provides an overview of the planned pharmacodynamic analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 10 Overview of Planned Biomarker Analyses

| Endpoint / Parameter/ | | Untransformed | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | | | A | Absolu | ite | Change from Baseline | | | | | | | |
| | Stat | Stats Analysis Summary Individual | | | | | | | lysis | Sum | Summary | | idual |
| | Т | T F L T F F L | | | | | Т | F | L | T | F | F | L |
| Biomarker - Part A: Healthy Subjects | | | | | | | | | | | | | |
| Percent inhibition of CD69 biomarker | | | | Υ | | Υ | | | | | | Υ | |
| Biomarker - Part C: Chronic Spontaneous Urticaria Subjects | | | | | | | | | | | | | |
| Percent Inhibition of CD69 biomarker | | | | Υ | | Υ | | | | | Υ | | |

# 9.2. Pharmacokinetics and Biomarker Analyses

A potential relationship between plasma exposures of GSK2646264 ( $C_{min}$ ) and changes in biomarker levels and primary endpoints will be explored graphically by plotting their respective time course profiles and systemic exposure versus response profiles. The responsibility for conducting PK-PD analyses will be CPMS. These analyses will not be part of this SAP and will be reported separately.

### 10. REFERENCES

GlaxoSmithKline Document Number 2013N167482\_01 (Protocol Amendment – 02-10-DEC-2014): A randomised double blind (sponsor unblinded), single and repeat ascending dose First Time in Human study in healthy subjects, cold urticaria and chronic spontaneous urticaria subjects to investigate safety, tolerability, pharmacodynamics and pharmacokinetics of GSK2646264.

ICH E9, ICH HARMONISED TRIPARTITE GUIDELINE 1998 http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E9/Step4/E9 Guideline.pdf

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol |
| | Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 11.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 11.7 | Appendix 7: Examination of Covariates and Subgroups |
| Section 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 11.10 | Appendix 10: List of Data Displays |
| Section 11.11 | Appendix 11: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 11.1.1. Protocol Deviation Definitions for Exclusion from predefined Populations

- Exclusions from the Study Populations should be defined prior to unblinding and should be summarized and listed [ICH E9, 1998, Section 5.2.2.] This will be included in Section 6.1 Study Populations.
  - Exclusions from study populations may be defined as a subset of the Important Deviations as appropriate. These details should be documented in the Plan for Managing Protocol Deviations and in the RAP.
  - Any planned exclusions from study populations which are not considered to be deviations, should be defined in the RAP with rationale and any programming details as appropriate.

## 11.1.2. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Failure of any inclusion/exclusion criteria |
| 02 | <ul> <li>Subjects who developed the withdrawal criteria but were not withdrawn</li> </ul> |
| 03 | Any deviation that impact the safety of subjects |
| 04 | Failed to provide scheduled assessment |
| 05 | Major deviation from the conduct of trial |

Protocol deviation definition criteria and resulting exclusion from analysis populations will be agreed and summarized in a separate protocol deviation definition document that has to be updated and reviewed on a regular basis.

# 11.2. Appendix 2: Time & Events

# 11.2.1. Protocol Defined Time & Events

# 11.2.1.1. Part A, Dose Group 1 (Healthy Volunteers)

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 | | | | | | Day 5 to Day<br>7 | |
| Admission to Unit | | Х | | | | | | |
| Informed Consent | Χ | | | | | | | |
| Demographics | Χ | | | | | | | |
| Complete physical | Χ | | | | | | X | |
| Body weight (kg) | Χ | | | | | | | |
| Height (cm) without | Х | | | | | | | |
| shoes | ^ | | | | | | | |
| Brief physical | | Χ | | | | | | |
| Medical/medication/drug/<br>alcohol history | Χ | | | | | | | |
| 12-lead ECG <sup>1</sup> | Χ | Х | | | | X | Х | Triplicate ECG at screening and CV risk factors questionnaire |
| Vital signs | Χ | Χ | Х | Χ | Χ | X | X | |
| Urine drug/alcohol screen | Χ | Х | | | | | | |
| HIV, Hep B and Hep C screen | Х | | | | | | | |
| Clinical Laboratory Tests | Χ | Х | | | | X | Х | |

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 | | | | | | Day 5 to Day<br>7 | |
| Allergen Challenge-<br>Skin Prick Test | X3,4 | | <b>X</b> 3, 5 | | X3,5 | X <sup>7</sup> | | 3. SPT- Skin Prick Test analysis will be performed at ~15-20mins post challenge. 4. SPT with all 4 specified allergens 5. SPT using one allergen will be performed 6 hours post dose (see Clinical Trial Protocol Section 6.4.1) 7. SPT using one allergen will be performed 24 hrs after the last dose |
| TSH <sup>2</sup> | Χ | | | | | | | 2. TSH test only at screening only |
| Randomisation | | Х | | | | | | |
| Tolerability Assessment | | | | $X_{8}$ | ← | → | | 9. Tolerability assessment at pre – and ~6 hours post-dose Note: No tolerability assessment on day 4. |
| AE assessment | | Х | | <b>←</b> | | | Х | |
| Concomitant Medication | | X | | <del></del> | | <del>-</del> | X | |
| Pharmacokinetic<br>Blood Sample <sup>6</sup> | | | Х | Х | Х | X8 | | 6.PK blood sample taken at pre<br>dose, 1,2, 4, 8, 12 and 24hr post<br>dose<br>8.PK refers to sample 24 hours<br>post dose |
| Study Treatment Dosing | | | X | Χ | Χ | | | |
| Discharge from unit | | | | | | X | | |
| Outpatient visit | Χ | | | | | | X | |

# 11.2.1.2. Part A: Healthy Volunteer Time and Event Table Dose group 2

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 | | | | | | | | | | Day 9 – Day<br>11 | |
| Admission to Unit | | Х | | | | | | | | | | |
| Informed Consent | Χ | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Complete physical | Х | | | | | | | | | | Х | |
| Body weight (kg) | Χ | | | | | | | | | | | |
| Height (cm) without shoes | Χ | | | | | | | | | | | |
| Brief physical | | Χ | | | | | | | | | | |
| Medical/medication/drug /alcohol history | Χ | | | | | | | | | | | |
| 12-lead ECG <sup>1</sup> | Х | Х | | | | | | | | Х | Х | Triplicate ECG at screening and CV risk factors questionnaire |
| Vital signs | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | |
| Urine drug/alcohol screen | Х | Χ | | | | | | | | | | |
| Urine for metabolite analysis | | | X10 | | | X <sup>22</sup> | | | | | | 10. Pre dose and pool samples taken 0-12 and 12-24 hours post dose 22. Pool samples taken 0-12 and 12-24 hours post |
| HIV, Hep B and Hep C screen | Х | | | | | | | | | | | |
| Clinical Laboratory Tests | X <sup>17</sup> | X <sup>17</sup> | | Xa | | Xa | X <sup>17</sup> | | X <sup>17</sup> | | X <sup>17</sup> | 9. Pre-dose AST, ALT, Alkaline Phosphatase, Total Bilirubin Only-: results to be communicated to the GSK Medical monitor on the same day 17.Clinical lab test as per Section 6.3.4 of the protocol |

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 | | | | | | | | | | Day 9 – Day<br>11 | |
| Allergen Challenge-<br>Skin Prick Test | X <sup>3,4</sup> | | X3,5 | | X <sup>3,5</sup> | X <sup>3,</sup> 5 | | X 3,7 | | | | 3. SPT- Skin Prick Test measurements will be performed ~15-20 mins post challenge. 4. SPT with all 4 specified allergens 5. SPT will be performed 6 hours post dose 7. SPT will be performed 48 hours post dose of Day 4 (on the morning of Day 6) |
| TSH <sup>2</sup> | Χ | | | | | | | | | | | 2. TSH test only at screening only |
| Randomisation | | Х | | | | | | | | | | |
| Tolerability Assessment | | | X <sup>11</sup> ← | | | | | | | | | 11. Tolerability assessment at pre – and ~6 hours post-dose on dosing days |
| AE assessment | | Х | | <b>←</b> | | | | | <del>-</del> | | Х | |
| Concomitant Medication | | Х | | <b>←</b> | | | | | <del>-</del> | | Х | |
| Pharmacokinetic<br>Blood Sample | | | Xe | Xe | Xe | X <sub>6</sub> | X <sup>18</sup> | X <sup>19</sup> | X <sup>20</sup> | X <sup>21</sup> | | 6. PK blood sample taken at pre dose, 1, 2, 4, 8, 12 and 24hours post previous dose 18. PK blood sample taken at 30, 36, 48 hours, post dose of Day 4 19. PK blood sample taken at 54, 60, 72 hours, post dose of Day 4 20. PK blood sample taken at 78, 84 hours post dose of Day 4 21. PK blood sample taken at 96 hours post dose of Day 4 |

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 | | | | | | | | | | Day 9 – Day<br>11 | |
| Blood Sample for CD69 expression | | | X12 | | | X <sup>13</sup> | X <sup>14</sup> | | X <sup>15</sup> | X <sup>16</sup> | | 12. Predose 13. 4 hours post dose of Day 4 14. 24 hours post dose of Day 4 (sample taken in the morning of day 5) 15. 72 hours post dose of Day 4 16. 96 hours post dose of Day 4 |
| Study Treatment Dosing <sup>8</sup> | | | Х | Х | Х | Х | | | | | | 8. This will be once daily dosing using fresh bottles at 1% strength in the morning |
| Discharge from unit | | | | | | | | | | Χ | | |
| Outpatient visit | X | | | | | | | | | | X | |

# 11.2.1.3. Part B (Cold Urticaria Subjects)

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7<br>days | | | | | | Day 5 to<br>Day 7 after<br>last dose | |
| Admission to Unit | | Χ | | | | | | |
| Informed Consent | Х | | | | | | | |
| Demographics | Х | | | | | | | |
| Complete physical | Х | | | | | | Х | |
| Body weight (kg) | X | | | | | | | |
| Height (cm) without shoes | Х | | | | | | | |
| Brief physical | | Х | | | | | | |
| Medical/medication/<br>drug/alcohol history | Х | | | | | | | |

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7<br>days | | | | | | Day 5 to<br>Day 7 after<br>last dose | |
| 12-lead ECG <sup>1</sup> | Х | Х | | | Х | | Х | Triplicate ECG at screening and CV risk factors questionnaire |
| Vital signs | Χ | Х | Х | Х | Х | | Х | |
| Urine drug/alcohol screen | Х | Х | | | | | | |
| Pregnancy Test (women) <sup>2</sup> | X(S) | | X(S/U) | | | | X(S) | 2. Pregnancy test will be performed 3 times during screening, serum on day -28, day -7 to -4, and a serum or urine pregnancy test the day of the start of the study prior to dosing and a serum pregnancy test at the follow up visit |
| HIV, Hep B and Hep C screen | Х | | | | | | | |
| Clinical Laboratory Tests | Х | Χ | | | Х | | Х | |
| Allergen Challenge- SPT | X4,5 | | X4,6 | | X4,6 | | | 4. SPT- Skin Prick Test measurements will be performed ~15-20mins post challenge 5. SPT using all 4 specified allergens 6. SPT will be performed at 6 hours post dose (see Clinical Trial Protocol Section 6.4.1) |
| TSH <sup>3</sup> | Х | | | | | | | 3. TSH test only at screening only |
| Cold Temp Test (Temp<br>Test 4.0) | Х | | Х | | Х | <b>X</b> <sup>7</sup> | | 7. 24 hours after last dose |
| Review of eligibility criteria and medication prior to randomisation | | Х | | | | | | |
| Randomisation | | Χ | | | | | | |
| Tolerability Assessment | | | X¹0 ← | | | | | 10. Tolerability assessment at pre – and ~6 hours post-dose |
| AE assessment | | Χ | ← | | | • | Х | |
| Concomitant Medication | | Х | | <del></del> | <del>-)</del> | <u> </u> | Х | |

| Day: | Screening | -1 | 1 | 2 | 3 | 4 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7<br>days | | | | | | Day 5 to<br>Day 7 after<br>last dose | |
| Pharmacokinetic Blood<br>Sample <sup>8</sup> | | | X | | Х | Xa | | <ul><li>8. PK blood sample taken at pre dose,1,2,4, 8, 12hr post dose</li><li>9. If only once daily dosing then a PK sample will be taken at 24h post dose</li></ul> |
| Study Treatment Dosing | | | Х | Х | Х | | | |
| Discharge from unit | | · | | | | Х | | |
| Outpatient visit | X | _ | | | | | X | |

# 11.2.1.4. Part C (Chronic Spontaneous Urticaria Cohort)

| Day: | Screening | 1 | 2 | 3 | 4 | 5 | 6 | 7 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 days | | | | | | | | 9-14 days after last dose | |
| Informed Consent | Х | | | | | | | | | |
| Demographics | Χ | | | | | | | | | |
| Complete physical | Χ | | | | | | | | Χ | |
| Body weight (kg) | Χ | | | | | | | | | |
| Height (cm) without shoes | Χ | | | | | | | | | |
| Brief physical | | Χ | | | | | | | Χ | |
| Medical/medication/<br>drug/alcohol history | Χ | | | | | | | | | |
| 12-lead ECG <sup>1</sup> | Х | Х | | | | | | Х | X | Triplicate ECG at screening and CV risk factors questionnaire |
| Vital signs | Х | Х | | | Χ | | | Χ | X | |
| Urine drug/alcohol screen | Х | Х | | | | | | | | |

| Day: | Screening | 1 | 2 | 3 | 4 | 5 | 6 | 7 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 days | | | | | | | | 9-14 days after last dose | |
| Pregnancy Test (women) <sup>2</sup> | X(S) | X<br>(S/U) | | | | | | | X(S) | 2. Pregnancy test will be performed 3 times during screening, serum (S) on day -28, day -7 to -4, and a serum or urine (U) pregnancy test the day of the start of the study prior to dosing and a serum pregnancy test at the follow up visit |
| HIV, Hep B and Hep C screen | Х | | | | | | | | | |
| Clinical Laboratory Tests | Χ | Χ | | | | | | Χ | Χ | |
| TSH <sup>3</sup> | Χ | | | | | | | | | 3. TSH test only at screening only |
| Blood Sample for CD69 expression <sup>11</sup> | | X <sub>9</sub> | | | | | | X <sup>10</sup> | | 9. Predose 10. 4 hours post dose 11 A decision will be made after Part A on whether samples are taken in Part C |
| Randomisation | | Χ | | | | | | | | |
| UAS-7 Diary⁴ | X | х | X | X | x | x | x | X | | 4. Screening UAS7 diary will be completed using 7 successive days before randomisation (day 1). If there is a lapse in any day prior to day 1 the subject must complete the full 7 days worth of diary entries again during the screening period. |
| QOL (DLQI) | Х | Χ | | | | | | Χ | | |
| AAS | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | |
| AE assessment | | X8 <b>←</b> | | | | | | -> | Х | Tolerability assessment at pre and post-dose |

| Day: | Screening | 1 | 2 | 3 | 4 | 5 | 6 | 7 | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (relative to Day 1) | -28 to -7 days | | | | | | | | 9-14 days after last dose | |
| BHR- Basophil Histamine Release<br>Test | | <b>X</b> 5 | | | | | | | | 5. Sample taken predose |
| Pharmacokinetic Blood Sample <sup>6</sup> | | Х | | | Х | | | Х | | 6. PK blood sample taken at predose sample and 2 and 4hr post dose |
| Study Treatment Dosing | | Х | X <sup>7</sup> | <b>X</b> <sup>7</sup> | Χ | <b>X</b> <sup>7</sup> | <b>X</b> <sup>7</sup> | Х | | 7. The nurse will visit the subject at home to apply the dose |
| Outpatient visit | Χ | Х | | | Χ | | | Χ | X | |

# 11.3. Appendix 3: Data Display Standards & Handling Conventions

#### 11.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| Α | GSK2646264 X.X mg | GSKX.X mg | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

In accordance with the body surface area (BSA) to be used Arm, Leg and Front Torso of the subjects had to be treated on the different body sides with either GSK2646264 or matching placebo treatment as displayed below:

Table 11 Overview of Treatments Doses and Analyses.

| Part | Dose | BSA<br>treated per<br>body side<br>(left/right) | Day<br>of Treatment<br>(Tests<br>performed) | Comment |
|---|---|---|---|---|
| А | 0.5%<br>(Group 1) | 0.2%<br>1%<br>5% | D1 (PK/PD)<br>D2 (PK)<br>D3 (PK/PD) | qd |
| A | 1.0%<br>(Group 2) | 5%<br>5%<br>10%<br>10% | D1 (PK/PD)<br>D2 (PK)<br>D3 (PK/PD)<br>D4 (PK) | qd |
| В | .0.5 or 1% | 0.2%+5%<br>0.2%+5%<br>0.2%+5% | D1(PK/PD)<br>D2<br>D3(PK/PD) | qd or bid<br>(D3 morning<br>dose only) |
| С | .0.5 or 1% | X.X2% | D1 (PK/PD) | Qd or bid |

maximum tolerated dose (taken from Part A)

<sup>1.</sup> Order represents treatments being presented in TFL. Placebo is to be presented at start in Tables, Figures and Listings. Dosing of GSK treatment will be displayed in ascending order, where appropriate.

<sup>&</sup>lt;sup>2</sup> maximum BSA treated (taken from Part A)

The following changes to treatment dosing were made to dose group 2 (Part A) in light of dose escalation review meeting at the end of dose group 1:

Table 12 Treatment applied to specified areas per day on Part A; healthy subjects, n=9, dose group 2

| | Day 1-2 | Day 3-4 | Day 5 to 7 |
|---|---|---|---|
| Area | <b>AM</b> <sup>a</sup> | AM <sup>a</sup> | |
| Left<br>Arm | 0.36g of 1.0%b GSK2646264 or placeb | NO<br>DOSING | |
| Right<br>Arm | 0.36g of 1.0% GSK2646264 or placebo | NO<br>DOSING | |
| Left | 9g of 1.0% b GSK2646264 or placebo | 18g of 1.0% b GSK2646264 or placebo | NO |
| Front | cream applied to 900cm <sup>2</sup> (~5% BSA) | applied to 1800cm <sup>2</sup> (~10% BSA) | DOSING |
| Torso | | | |
| Right | 9g of 1.0% b GSK2646264 or placebo | 18g of 1.0% b GSK2646264 or placebo | NO |
| Front | applied to 900cm <sup>2</sup> (~5% BSA) | applied to 1800cm² (~10% BSA) | DOSING |
| Torso | | | |

a. AM dosing only

#### 11.3.2. Baseline Definition & Derivations

#### 11.3.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Parameter Study Assessments Considered As Baseline | | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety Assessment | | | | |
| Laboratory | X | <b>X</b> <sup>2</sup> | | Day -1,<br>(Part A & B)<br>Screening (Part C) |
| Vital Signs | Х | | X | Day 1 (pre) |
| ECG | Х | Х | | Screening <sup>1</sup> |
| Pharmacodynamics | | | | |
| Allergen Challenge<br>SPT (Part A & B) | | | | No baseline |
| Cold Temp test<br>(Part B) | | | | No baseline |
| UAS7 (Part C) | Х | | | Screening |
| AAS (Part C) | Х | | | Screening |

b. 0.5% strength may be used if data for Part A and/or group 2 supports
| Parameter | Study Assessments Considered As Baseline | | | Baseline Used in |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Health Outcome | | | | |
| DLQI (Part C) | X | | | Screening |

#### NOTES:

- 1. Use the mean of replicate assessments at any given time point as the value for that time point in all summaries, figures and statistical analyses.
- 2. Not in Part C

### 11.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| % inhibition | =[(control – treatment)/control]x100 |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.3.2.1 Baseline Definitions will be
  used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- As only one baseline will be defined for all parameters (i.e. at the start of the study), there will only be one baseline on all summaries (i.e. not a separate baseline for each subsequent repeat dose).
- The baseline definition will be footnoted on all change from baseline outputs, where applicable.
- If baseline value for (day -1) is missing, screening value will be used as baseline. If both assessments are missing then no derivation will be performed and will be set to missing.

### 11.3.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | |
| , | oported versions of SAS software will be used to perform all data analyses and plays (tables, figures, and listings). |
| Reporting Area | |
| HARP Server | PHU058 |
| HARP Area | : \ARWORK\GSK2646264\final or \ARWORK\GSK2646264\final |
| QC Spreadsheet | : Not applicable ] |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC / ADaM Standards Library standards. For<br/>creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be<br/>implemented for conversion from SI to SDTM.</li> </ul> | |
| Generation of Files | |
| PDF files will be generated. | |

### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

### **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| | N, n, mean, 95% CI of the mean, standard deviation (SD), median, |
| | minimum (min) and maximum (max). |
| Categorical Data | N, n, frequency, % |

### **Reporting of Pharmacokinetic Concentration Data**

| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

#### Reporting of Pharmacokinetic Parameters

| Descriptive | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) |
|---|---|
| Summary Statistics | of logged data and [between and or within] geometric coefficient of variation |

| Reporting Standards | |
|---|---|
| (Log Transformed) | (CVb/w (%)) will be reported. |
| | [1] $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of log transformed data) |
| | [2] $CV_w$ (%) = $\sqrt{(exp(MSE) - 1) * 100}$ |
| | (MSE = mean square error from mixed effect model of loge-transformed data). |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 11.4. Appendix 4: Derived and Transformed Data

### 11.4.1. General

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing → Study Day = Missing
  - Randomisation Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

### 11.4.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 11.4.3. Safety

### **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTeF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}} \qquad \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

| Adverse Events | |
|---|---|
| AE Type | Derivations |
| AE Onset Time | ➤ If Treatment Start Date > AE Onset Date : |
| Since First Dose | = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date ≤ AE Onset Date : |
| | = AE Onset Date - Treatment Start Date + 1 |
| | Missing otherwise |
| AE Duration (Days) | > AE Resolution Date – AE Onset Date + 1 |
| AE = On Treatment | If AE onset date is on or after the treatment start date and on or<br>before the treatment stop date. |
| AE = Post Treatment | ➤ If AE onset date is after the treatment stop date. |
| AE = Drug-related | ➢ If relationship is marked 'YES' on eCRF OR value is missing. |
| Current update | |
| MedRA version | |
| 17.1 will be used | |

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

### **Tolerability Assessments**

Tolerability will be assessed with the skin irritation scoring system for Part A and B of study, where the score consists of a numeric score according to the dermal response scoring i), and a letter according to the other effects scoring ii), as follows

- 0 =no evidence of irritation
- 1 = minimal erythema, barely perceptible (pink)
- 2 = moderate erythema (definite redness), readily visible; minimal edema or minimal papular response
- 3 = strong erythema (intense redness), or erythema and papules
- 4 = definite edema
- 5 = erythema, edema, and papules
- 6 = vesicular eruption
- 7 = strong reaction spreading beyond test site
- ii) Other effects:
- Z = no other effect
- A =slight glazed appearance
- B = marked glazing
- C = glazing with peeling and cracking
- F = glazing with fissures
- G = film of dried serous exudate covering all or part of the patch site
- H = small petechial erosions and/or scabs

For each skin assessment, letter grade will be converted to numeric values as below: A=0,Z=0, B=1, C=2, F=3, G=3, H=3. A combined score for each subject will be calculated by adding all numeric and letter scores. A maximum score of 3 is allowed. Mean irritation score for each subject will be computed through the study period. Mean score will be analyzed.

# 11.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

### 11.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as subjects who completed all visits of the study including the follow-up visit.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 11.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: The collection instrument Collection Collection |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not<br/>considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any subjects excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |
| UAS7 score | In presence of one or more missing daily UAS7 scores, the following algorithm will be applied: |
| | <ul> <li>If a patient has at least 4 non-missing daily UAS7 scores within the 7 days,<br/>the UAS7 score will be calculated as the sum of the available eDiary UAS7<br/>scores in that week, divided by the number of days that have a non-missing<br/>diary UAS7 score, multiplied by 7.</li> </ul> |
| | <ul> <li>If there are less than 4 non-missing daily UAS7 scores, then the UAS7 score<br/>will be missing.</li> </ul> |
| AAS | Missing values will not be imputed |
| DLQI | 1. If one question is left unanswered this is scored 0 and the scores are summed and expressed as usual out of a maximum of 30. |
| | 2. If two or more questions are left unanswered the questionnaire is not scored. |
| | 3. If question 7 is answered 'yes' this is scored 3. If question 7 is answered 'no' or |
| | 'not relevant' but then either 'a lot' or 'a little' is ticked this is then scored 2 or 1. If it is answered 'no', but the second half is left incomplete, the score will remain 0. |
| | 4. If two or more response options are ticked, the response option with the highest score should be recorded. |
| | 5. If there is a response between two tick boxes, the lower of the two score options |

| Element | Reporting Detail |
|---|---|
| | should be recorded. |
| | 6. When using sub-scales, if the answer to one question in a sub-scale is missing, |
| | that sub-scale should not be scored. |

# 11.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

### 11.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.6. Appendix 6: Values of Potential Clinical Importance

# 11.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓ 0.075 | |
| | ,, | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓ 25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |
| Red Blood Cell Count (RBC) | x10 <sup>6</sup><br>cells/µL | | 4.2 | 5.9 |
| Mean Corpuscular Volume (MCV) | fL | | 80 | 100 |
| Mean Corpuscular Hemoglobin (MCH) | pg | | 28 | 32 |
| Mean Corpuscular Hemoglobin Concentration (MCHC) | g/L | | 32 | 36 |
| Monocytes | x10 <sup>9</sup> / L | | | 0.208 |
| Eosinophils | x10 <sup>9</sup> / L | | | 0.44 |
| Basophils | x10 <sup>9</sup> / L | | | 0.01 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| | mmol/L | | | 1.3*ULN |
| Creatinine | µmol/L | | | 159 |
| | µmol/L | $\Delta$ from BL | | 44 |
| Glucose | mmol/L | | 3 | 11.1 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|----------------|-------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |

| Liver Function | | | |
|-------------------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 1.5x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |
| Urea Nitrogen (BUN) | mmol/L | Low | <2.9 |
| Urea Nitrogen (BUN) | mmol/L | High | >7.1 |
| Chloride | mmol/L | Low | <98 |
| Chloride | mmol/L | High | >106 |
| Gamma-glutamyl Transpeptidase | U/L | Low | <8 |
| (GGT) | U/L | High | >78 |
| Direct Bilirubin | µmol/L | High | >5.1 |
| Total Protein | g/L | Low | <60 |
| TOTAL FIOLEIT | g/L | High | >78 |

# 11.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | • | | |
| Abaduta OTa Intanial | msec | > 450 [2] | ≤ 479 <sup>[2]</sup> |
| Absolute QTc Interval | | ≥ 480 <sup>[2]</sup> | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 [ | > 110 |
| Change from Baseline | | | |
| | msec | > 60 | |
| Increase from Baseline QTc | msec | > 30 | ≤ 59 |
| | msec | ≥ 60 [ | |

# 11.6.3. Vital Signs

| Vital Sign Parameter Units | | Clinical Concern Range | |
|----------------------------|------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |


| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

# 11.7. Appendix 7: Examination of Covariates, Subgroups & Other Strata

# 11.7.1. Handling of Covariates, Subgroups & Other Strata

• Not applicable.

# 11.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

# 11.8.1. Statistical Analysis Assumptions

| Endpoint(s) | PD Parameters |
|---|---|
| Analysis | <ul> <li>ANOVA to estimate the effect of GSK2646264 relative to Placebo as<br/>comparison of interest. Point estimates and corresponding 95% confidence<br/>intervals will be constructed.</li> </ul> |
| Analysis | ANCOVA. |
| | <ul> <li>Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.</li> <li>If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.</li> </ul> |
| Analysis | Logistic Regression |
| | <ul> <li>Model fit will be assesses by</li> <li>plotting observed probability vs predictive probability</li> <li>Chi-square test for goodness fit test</li> </ul> |

# 11.9. Appendix 9: Abbreviations & Trade Marks

# 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AAS | Angioedema Activity Score |
| AE | Adverse Event |
| ALT | Alanine aminotransferase (SGPT) |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) |
| . , | extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to |
| | last time of quantifiable concentration |
| $AUC(0-\tau)$ | Area under the concentration-time curve over the dosing interval |
| BHR | Basophil Histamine Release |
| BMI | Body mass index |
| BP | Blood pressure |
| BPM | Beat Per Minute |
| BQL | Below the quantification limit |
| BUN | Blood urea nitrogen |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPDS | Clinical Pharmacology Data Sciences |
| CPK | Creatine phosphokinase |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CsU | Chronic spontaneous Urticaria |
| CU | Cold Urticaria |
| CV | Coefficient of variance |
| DBP | Diastolic blood pressure |
| ECG | Electrocardiogram |
| FTIH | First time in humans |
| GGT | Gamma glutamyltransferase |
| GSK | GlaxoSmithKline |
| hCG | Human chorionic gonadotropin |
| HIV | Human Immunodeficiency Virus |
| h/hr | Hour(s) |
| HR | Heart rate |
| IP | Investigational Product |
| IU | International Unit |
| Kg | Kilogram |
| $\lambda z$ | Terminal phase rate constant |
| L | Liter |
| ln | Naperian (natural) logarithm |

| Abbreviation | Description |
|--------------|------------------------------------------------------|
| LOQ | Limit of quantification |
| LLQ | Lower limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligrams |
| mL | Milliliter |
| msec | Milliseconds |
| NQ | Non-quantifiable concentration measured as below LLQ |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| QD | Once daily |
| RAP | Reporting and Analysis Plan |
| RBC | Red blood cells |
| SAE | Serious adverse event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SUSAR | Suspected, Unexpected, Serious Adverse drug Reaction |
| t½ | Terminal phase half-life |
| τ | Dosing interval |
| tmax | Time of occurrence of Cmax |
| ULN | Upper limit of normal |
| WBC | White blood cells |
| GSK | GlaxoSmithKline |

### 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| SAS/STAT |

### 11.10. Appendix 10: List of Data Displays

### 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|----------------|
| Study Population | 1.1 to 1.8 | Not applicable |
| Safety | 3.1 to 3.18 | Not applicable |
| Pharmacokinetic | 4.1 to 4.3 | 4.1 to 4.3 |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.15 | 5.1 to 5.14 |
| Section | List | ings |
| ICH Listings | 1 to 28 | |
| Other Listings | 29 t | o 35 |

### 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Other Listings | | | OTHER_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 11.10.3. Deliverable [Priority]

| | Delivery [Priority] [1] | Description |
|---|-------------------------|------------------------------------------------|
| Ī | IA [X] | Interim Analysis Statistical Analysis Complete |
| | SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 11.10.4. Study Population Tables

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Dispos | ition | | | | |
| 1.1. | Safety | CP_ES1 | Summary of Subject Disposition | Programmer to update primary reason for withdrawal to be study specific. Please only include Total column (not treatment columns) | IA[1], SAC [1] |
| 1.2. | Safety | SA1 | Summary of Study Populations | | IA[1],SAC [1] |
| 1.3. | Safety | DVA1 | Summary of Important Protocol Deviations | Generated, if data permits. As required, refer to PDMP. Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 1.4. | Safety | SD1 | Summary of Investigational Product Status | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| Demog | raphics | | | | |
| 1.5. | Safety | DM1 | Summary of Demographic Characteristics | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| Medica | l History | 1 | | , | ı |
| 1.7. | Safety | MH4 | Summary of Medical History | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| Concor | mitant Medicati | on | | | |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Safety | CP_CM1 | Summary of Concomitant Medications by Generic Term | Please only include Total column (not treatment columns) | IA[1],SAC [1] |

# 11.10.5. Efficacy Tables

Not applicable.

# 11.10.6. Safety Tables

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Drug E | xposure | | | | |
| 3.1. | Safety | EX1 | Summary of Exposure to Study Drug | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| Advers | e Events | | | | |
| 3.2. | Safety | CP_AE1p | Summary of All Adverse Events | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 3.3. | Safety | CP_AE1p | Summary of Drug-Related Adverse Events | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 3.4. | Safety | CP_AE1p | Summary of All Localised Adverse Events | | IA[1],SAC [1] |
| 3.5. | Safety | CP_AE1p | Summary of Serious Adverse Events | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 3.6. | Safety | CP_AE1p | Summary of AEs Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 3.7. | Safety | AE5 | Summary of Adverse Events by Maximum Intensity/Grade | Please only include Total column (not treatment columns) | IA[1],SAC [1] |
| 3.8. | Safety | AE2 | Relationship between System Organ Class and Verbatim Text | | IA[1],SAC [1] |
| Clinica | Laboratory As | ssessments | | | |
| 3.9. | Safety | LB1 | Summary (Absolute and Change from Baseline) of Clinical Chemistry Laboratory Values | Please only include Total column (not treatment columns). Order parameters alphabetically | IA[1],SAC [1] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | LB2 | Summary of Clinical Chemistry Data Outside the Reference Range | Order parameters alphabetically | IA[1],SAC [1] |
| 3.11. | Safety | LB1 | Summary (Absolute and Change from Baseline) of Haematology Laboratory Values | Please only include Total column (not treatment columns).Order parameters alphabetically | IA[1],SAC [1] |
| 3.12. | Safety | LB2 | Summary of Haematology Data Outside the Reference Range | Order parameters alphabetically | IA[1],SAC [1] |
| 3.13. | Safety | UR3 | Summary of Urinalysis Dipstick Results | Please only include Total column (not treatment columns).Order parameters alphabetically | IA[1],SAC [1] |
| Electro | cardiogram (EC | CG) | | | |
| 3.14. | Safety | EG1 | Summary (Absolute and Change from Baseline) of ECG Findings | Please only include Total column (not treatment columns).Order parameters alphabetically | IA[1],SAC [1] |
| 3.15. | Safety | EG2 | Summary (Absolute and Change from Baseline) of ECG Values | Please only include Total column (not treatment columns).Order parameters alphabetically | IA[1],SAC [1] |
| Vital Si | gns | | | | |
| 3.16. | Safety | VS1 | Summary (Absolute and Change from Baseline) of Vital Signs | Please only include Total column (not treatment columns).Order parameters alphabetically | IA[1],SAC [1] |
| Tolerab | Tolerability assessment | | | | |
| 3.17. | Safety | Non- Standard<br>SAFE_T1 | Summary (Absolute and Change from Baseline) of Mean irritation score assessment | | IA[1],SAC [1] |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.18. | Safety | Non- Standard<br>SAFE_T2 | Assessment of Maximum Dermal Reactions and Response | | IA[1],SAC [1] |


200196

# 11.10.7. Safety Figures

Not applicable.

### 11.10.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetics | | | | |
| 4.1. | PK | PKCT1 | Summary of Serum GSK2646264 Pharmacokinetic Concentrations versus time by actual dose | | IA[1],SAC [1] |
| 4.2. | PK | PKPT1 | Summary of Derived Serum GSK2646264 Pharmacokinetic Parameters by actual dose | | IA[1],SAC [1] |
| 4.3. | PK | PKPT3 | Summary of Log-Transformed Derived Serum GSK2646264 Pharmacokinetic Parameters by actual dose | | IA[1],SAC [1] |

# 11.10.9. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetics | | | | |
| 4.1. | PK | PKCF1 | Individual Serum GSK2646264 Concentration-Time Plot (Linear and Semi-log) | x-axis should display Actual relative time Include line for LLQ along with footnote defining LLQ value. Include values below LLQ | IA[1],SAC [1] |
| 4.2. | PK | PKCF3 | Median Serum GSK2646264 Concentration-Time Plot (Linear and Semi-log) | X-axis should display Planned relative time Include line for LLQ along with footnote defining LLQ value. Include values below LLQ Use different symbols for treatments | IA[1],SAC [1] |
| 4.3. | PK | PKCF4 | Mean and SD of Serum GSK2646264 Concentration-Time Plot (Liner and Semi-log) | X-axis should display Planned relative time Include line for LLQ along with footnote defining LLQ value. Include values below LLQ Use different symbols for treatments | IA[1],SAC [1] |

# 11.10.10. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acodynamics | | | | |
| 5.1. | PD | Non-<br>Standard_PDT<br>1 | Allergen Challenge, Weal Area - Summary Statistics (Absolute and Percent of Inhibition) | Absolute and Percent of Inhibition Part A + B | IA[1],SAC [1] |
| 5.2. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Allergen Challenge, Weal Volume – Summary Statistics (Absolute and Percent of Inhibition) | Absolute and Percent of Inhibition Part A + B | IA[1],SAC [1] |
| 5.3. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Allergen Challenge, Longest Weal Diameter- Summary Statistics (Absolute and Percent of Inhibition) | Absolute and Percent of Inhibition Part A + B | IA[1],SAC [1] |
| 5.4. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Allergen Challenge, Weal perpendicular length - Summary Statistics (Absolute and Percent of Inhibition) | Absolute and Percent of Inhibition Part A + B | IA[1],SAC [1] |
| 5.5. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Allergen Challenge, Flare Erythema - Summary Statistics (Absolute and Percent of Inhibition) | Absolute and Percent of Inhibition Part A + B | IA[1],SAC [1] |

| Pharma | acodynamic an | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Cold Temp Test, Change in critical temperature thresholds | Absolute<br>Part B only | SAC [1] |
| 5.7. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | UAS7 Scores – Summary Statistics (Absolute and Change from Baseline) | Absolute and Change from Baseline Part C only | SAC [1] |
| 5.8. | PD | Example Non-<br>Standard_PDT<br>2 | Change from baseline in composite total UAS7 Scores – Treatment Comparison | Paired t-Test (95%CI) and ANCOVA to compare treatments groups. Pre-Dose Value as Covariate Part C only | SAC [1] |
| 5.9. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | UAS7 Components – Summary Statistics (Absolute and Change from Baseline) | Absolute and Change from Baseline<br>Part C only | SAC [1] |
| 5.10. | PD | Example Non-<br>Standard_PDT<br>2 modified<br>based on<br>endpoint. | Change from baseline in composite total UAS7 Components – Treatment Comparison | Paired t-Test (95%CI) and ANCOVA to compare treatments groups. Pre-Dose Value as Covariate Part C only | SAC [1] |

| Pharma | codynamic an | d Biomarker: Tab | les | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.11. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Angioedema Activity Score (AAS) – Summary Statistics (Absolute and Change from Baseline) | Absolute and Change from Baseline Part C only | SAC [1] |
| 5.12. | PD | Example Non-<br>Standard_PDT<br>2 modified<br>based on<br>endpoint. | Change from baseline in total Angioedema Activity Score (AAS) – Treatment Comparison | Paired t-Test (95%CI) and ANCOVA to compare treatments groups. Pre-Dose Value as Covariate Part C only | SAC [1] |
| 5.13. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Dermatology Life Quality Index (DLQI) – Summary Statistics (Absolute and Change from Baseline) | Absolute and Change from Baseline<br>Part C only<br>Sum-Score and Analysis of<br>Subscores | SAC [1] |
| 5.14. | PD | Example Non-<br>Standard_PDT<br>2 modified<br>based on<br>endpoint. | Change from baseline in total Dermatology Life Quality Index (DLQI) – Comparison Improvement from baseline | Paired t-Test (95%CI) Part C only No treatment comparison involved. Improvement from baseline in Quality Index | SAC [1] |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Biomar | ker | | | | |
| 5.15. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Inhibition of CD69 biomarker by strength, BSA and day – Summary Statistics | Part A + C | IA[1],SAC [2] |
| 5.16. | PD | Example Non-<br>Standard_PDT<br>1 modified<br>based on<br>endpoint. | Relationship between Basophil Histamine (BHR) test and Weal Characteristics | Part C only No treatment comparison involved. | SAC[2] |

# 11.10.11. Pharmacodynamic Figures

| Pharma | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | codynamics | | | | |
| 5.1. | PD | Non-Standard<br>_PD_F1 | Allergen Challenge, Weal Area (Percent of Inhibition) - Individual Subject Plot | Part A + B Page by : Treatment X-Axis : Continuous scale for visit (days) Y-Axis : Scaled accordingly to Parameter and include parameter name Legend : Subject | SAC [1] |
| 5.2. | PD | Non-Standard<br>_PD_F2 | Allergen Challenge, Weal Area (Percent of Inhibition, absolute value) - Box Plot | Part A + B X-Axis : Days Y-Axis : Result Legend : Treatment | SAC [1] |

| | No Population IDSL/TST ID / Title | | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.3. | PD | Example Non-<br>Standard<br>_PD_F1 | Allergen Challenge, Weal Volume (Percent of Inhibition) - Individual Subject Plot | Part A + B Page by : Treatment X-Axis : Continuous scale for visit (days) Y-Axis : Scaled accordingly to Parameter and include parameter name Legend : Subject | SAC [1] |

| Pharma | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.4. | PD | Example Non-<br>Standard<br>_PD_F2 | Allergen Challenge, Weal Volume (Percent of Inhibition, absolute value) - Box Plot | Part A + B X-Axis : Days Y-Axis : Result Legend : Treatment | SAC [1] |
| 5.5. | PD | Example Non-<br>Standard<br>_PD_F1 | Allergen Challenge, longest weal Diameter (Percent of Inhibition) - Individual Subject Plot | Part A + B Page by : Treatment X-Axis : Continuous scale for visit (days) Y-Axis : Scaled accordingly to Parameter and include parameter name Legend : Subject | IA[1],SAC [1] |
| 5.6. | PD | Example Non-<br>Standard<br>_PD_F2 | Allergen Challenge, longest Weal Diameter (Percent of Inhibition, absolute value) - Box Plot | Part A + B X-Axis : Days Y-Axis : Result Legend : Treatment | IA[1],SAC [1] |

| Pharma | acodynamic : F | igures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.7. | PD | Example Non-<br>Standard<br>_PD_F1 | Allergen Challenge, Weal perpendicular length (Percent of Inhibition) - Individual Subject Plot | Part A + B Page by : Treatment X-Axis : Continuous scale for visit (days) Y-Axis : Scaled accordingly to Parameter and include parameter name Legend : Subject | IA[1],SAC [1] |
| 5.8. | PD | Example Non-<br>Standard<br>_PD_F2 | Allergen Challenge, Weal perpendicular length (Percent of Inhibition, absolute value) - Box Plot | Part A + B X-Axis : Days Y-Axis : Result Legend : Treatment | IA[1],SAC [1] |
| 5.9. | PD | Example Non-<br>Standard<br>_PD_F1 | Allergen Challenge, Flare Erythema (Percent of Inhibition) - Individual Subject Plot | Part A + B Page by : Treatment X-Axis : Continuous scale for visit (days) Y-Axis : Scaled accordingly to Parameter and include parameter name Legend : Subject | IA[1],SAC [1] |

| Pharma | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.10. | PD | Example Non-<br>Standard<br>_PD_F2 | Allergen Challenge, Flare Erythema (Percent of Inhibition, absolute value) - Box Plot | Part A + B X-Axis : Days Y-Axis : Result Legend : Treatment | IA[1],SAC [1] |
| 5.11. | PD | Example Non-<br>Standard<br>_PD_F1 | Cold Temp Test (Change) - Individual Subject Plot | Part B only Page by: Treatment X-Axis: Continuous scale for visit (days) Y-Axis: Scaled accordingly to Parameter and include parameter name Legend: Subject | SAC [1] |
| 5.12. | PD | Example Non-<br>Standard<br>_PD_F2 | Cold Temp Test (Change) - Mean (95% CI) Plot | Part B only X-Axis : Days Y-Axis : Mean (± 95% CI) Result Legend : Treatment | SAC [1] |
| 5.13. | PD | Example Non-<br>Standard<br>_PD_F2 | UAS7 Score (Change from Baseline) - Mean (95% CI) Plot | Part C only X-Axis : Days Y-Axis : Mean (± 95% CI) Result Legend : Treatment | ,SAC [1] |

| Pharma | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.14. | PD | Example Non-<br>Standard<br>_PD_F2 | Angiodema Activity ScoreScore (AAS) (Change from Baseline) - Mean (95% CI) Plot | Part C only X-Axis : Days Y-Axis : Mean (± 95% CI) Result Legend : Treatment | SAC [1] |
| 5.15. | PD | Example Non-<br>Standard<br>_PD_F2 | Dermatology Life Quality Index (DLQI) - Box Plot | Part C only X-Axis : Days Y-Axis : Result Legend : Treatment | SAC [1] |

# 11.10.12. ICH Listings

| ICH : Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Randor | Randomisation | | | | |
| 1. | Safety | CP_TA1 | Listing of Randomised and Actual Treatments | | IA [1], SAC [1] |
| Subject | Disposition | | | | |
| 2. | Safety | ES7 | Listing of Reasons for Screen Failure | | IA [1], SAC [1] |
| 3. | Safety | ES2 | Listing of Reasons for Withdrawal | | IA [1], SAC [1] |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | | IA (SAC) |
| 5. | Safety | ES2 | Listing of Exclusions from Per Protocol Population | | IA (SAC) |
| Inclusio | on and Exclusion | on Criteria | | | |
| 6. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | IA [1], SAC [1] |
| Demog | rahics | | | | |
| 7. | Safety | DM2 | Listing of Demographic Characteristics | | IA [1], SAC [1] |
| 8. | Safety | DM9 | Listing of Race | | IA [1], SAC [1] |
| Medica | l History | | | | |
| 9. | Safety | MH2 | Listing of Medical History | | IA [1], SAC [1] |
| Concor | Concomitant Medication | | | | |
| 10. | Safety | CP_CM3 | Listing of Concomitant Medication by Generic Term | | IA [1], SAC [1] |
| Study [ | Drug Exposure | | | | |
| 11. | Safety | EX3 | Listing of Exposure Data | If applicable adapt to study data | IA [1], SAC [1] |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 12. | Safety | AE7 | Listing of All Adverse Events | | IA [1], SAC [1] |
| 13. | Safety | CP_AE8 | Listing of Subject Numbers for Individual Adverse Events | | IA [1], SAC [1] |
| 14. | Safety | CP_AE8a | Listing of Serious Adverse Events | | IA [1], SAC [1] |
| 15. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | IA [1], SAC [1] |
| Clinica | Laboratory As | sessments | | | |
| 16. | Safety | CP_LB5 | Listing of Haematology Abnormalities of Potential Clinical Importance | | IA [1], SAC [1] |
| 17. | Safety | CP_LB5 | Listing of All Haematology Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance | Including change from Baseline | IA [1], SAC [1] |
| 18. | Safety | CP_LB5 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | | IA [1], SAC [1] |
| 19. | Safety | CP_LB5 | Listing of Clinical Chemistry Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance | Including change from Baseline | IA [1], SAC [1] |
| 20. | Safety | CP_LB5 | Listing of All Hematology Laboratory Data for Subjects with Adverse Events of Interest | | IA [1], SAC [1] |
| 21. | Safety | UR2b | Listing of Urinalysis Data for Subjects with Abnormalities of Potential Clinical Concern | | IA [1], SAC [1] |
| Electro | cardiogram (E | CG) | | | |
| 22. | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance | | IA [1], SAC [1] |
| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with a Value of Potential Clinical Importance | Including change from Baseline | IA [1], SAC [1] |
| 24. | Safety | CP_EG5 | Listing of Abnormal ECG Findings | | IA [1], SAC [1] |
| Vital Sig | gns | | | • | • |
| 25. | Safety | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance | | IA [1], SAC [1] |
| 26. | Safety | CP_EG3 | Listing of All Vital Sign for Subjects with a Value of Potential Clinical Importance | Including change from Baseline | IA [1], SAC [1] |
| 27. | Safety | CP_VS4 | Listing of All Vital Signs for Subjects with Values of Potential Clinical Importance | | IA [1], SAC [1] |

# 11.10.13. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Tolerak | ility assessme | nt | | • | |
| 28. | Safety | Non-<br>Standard_Other<br>_L1 | Listing of irritation score assessment | | IA [1], SAC [1] |
| Pharma | acokinetics | | | | |
| 29. | PD | pkcl1p | Listing of GSK2646264 plasma PK Concentration-Time Data | | IA[1],SAC [1] |
| 30. | PD | pkpl1p | Listing of derived GSK2646264 plasma PK parameters | | IA[1],SAC [1] |
| Pharma | acodynamics | | | | |
| 31. | PD | Non-Standard<br>_Other_L2 | Listing of Allergen Challenge Parameters | Absolute and percent of inhibition to be presented. Part A + B | IA[1],SAC [1] |
| 32. | PD | Example Non-<br>Standard<br>_Other_L2<br>modified based<br>on endpoint. | Listing of Critical Temperature Thresholds | Absolute and change from baseline result to be presented. Part B only | SAC [1] |
| 33. | PD | Example Non-<br>Standard<br>_Other_L2<br>modified based<br>on endpoint. | Listing of UAS7 Scores and Subscores | Absolute and change from baseline result to be presented. Part C only | SAC [1] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 34. | PD | Example Non-<br>Standard<br>_Other_L2<br>modified based<br>on endpoint. | Listing of Angioedema Activity Score(AAS) | Absolute and change from baseline result to be presented. Part C only | SAC [1] |
| 35. | PD | Example Non-<br>Standard<br>_Other_L2<br>modified based<br>on endpoint. | Listing of Dermatology Life Quality Index (DLQI) | Absolute and change from baseline result to be presented. Total score and Subscores Part C only | SAC [1] |

# 11.11. Appendix 11: Example Mock Shells for Data Displays

Example : Non- Standard\_SAFE\_T1 Page x of y

Protocol : 2013N167482\_01

Population : Safety

Table 3.17
Summary (Absolute and Change from Baseline) of Mean irritation score assessment

| Treatment | Visit | Mean Irritation<br>Score | Mean of change<br>from baseline<br>Irritation Score |
|---|---|---|---|
| GSK2646264 0.5% | XX | XX | XX |
| XXXX | XX | XX | XX |
| Placebo | xx | xx | xx |

Page x of y

Example : Non- Standard\_SAFE\_T2

: 2013N167482\_01

Population : Safety

Protocol

Table 3.18
Assessment of Maximum Dermal Reactions and Response

| | | | GSK2646264 | GSK2646264 | |
|---|---|---|---|---|---|
| | Reaction | | (0.5%) | (1.0%) | Placebo |
| Assessment | Grade | Statistic | (N = XX) | (N = XX) | (N = XX) |
| Dermal Response | 1 | n (%) | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| - | 2 | n (%) | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| | - | <del>-</del> | | | ` <b>-</b> |
| | _ | | | | |
| | 7 | n (%) | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| Any Dermal | | | | | |
| Reaction | | n (%) | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| Grade 3 reaction | | | | | |
| (the mean time to | | n (%)(mean | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| get Grade 3) | | time (days)) | (XX.XX) | (XX.XX) | (XX.XX) |
| score ≥3 on the | | | | | |
| dermal response | | | | | |
| grading scale or | | | | | |
| a letter score of | | | | | |
| F, G, or H for | | n (%)(mean | XX (XX.XX) | XX (XX.XX) | XX (XX.XX) |
| other effects | | time (days)) | (XX.XX) | (XX.XX) | (XX.XX) |
| | | , ± , , | , | | · |

N: Number of subjects dosed with each treatment; n: Number of subjects with adverse event with particular reaction grade; %: Calculated using the number of subjects treated with each treatment as the denominator (n/N\*100);

200196

Example : Non-Standard\_PD\_T1 Page 1 of X
Protocol : 2013N167482\_01

Population : PD

 Table 5.1

 Allergen challenge, Weal Area- Summary Statistics (Absolute and Percent of Inhibition)

## Summary: Absolute

| Treatment | Time | | | CI 95% | CI 95% | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | N | Mean | Lower | Upper | S.D | Min | Median | Max |
| Placebo | Χ | Х | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | x | xxx.x | XXX.X | XXX.X | xx.xx | XXX | XXX | XXX |
| | Χ | X | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| GSK2646264<br>(0.5%) | Χ | х | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | X | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | Х | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | | | | | • | | | | |
| GSK2646264 | | | | | | | | | |
| (1.0%) | Χ | X | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | Χ | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | Χ | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |

| Programming Notes : | [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table |
|---|---|
| | [2] If absolute and percent inhibition fit in one table results can be unified in one table. |


200196


Example : Non-Standard\_PD\_T1 (Continued)

Protocol : 2013N167482\_01

Population : PD

 Table 5.1

 Allergen challenge, Weal Area- Summary Statistics (Absolute and Percent of Inhibition)

Summary: Percent of Inhibition

| Treatment | Time | Time | | CI 95% | CI 95% | | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|
| | | N | Mean | Lower | Upper | S.D | | | |
| Placebo | Χ | Х | XXX.X | | | | | | |
| | Χ | Χ | XXX.X | | | | | | |
| | Χ | X | XXX.X | | | | | | |
| GSK2646264<br>(0.5%) | Х | х | XXX.X | XXX.X | XXX.X | xx.xx | XXX | XXX | XXX |
| | Χ | x | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | Χ | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | | • | | | • | • | | | |
| GSK2646264 | ., | | | | | | | | |
| (1.0%) | Χ | Χ | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | X | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| | Χ | X | XXX.X | XXX.X | XXX.X | XX.XX | XXX | XXX | XXX |
| ETC | | | | | | | | | |

| Programming Notes : | [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table |
|---|---|
| . rogramming motor . | [1] For applicable enapoints, metade parameter as officer as 2 parameter of as more column in the table |
| | [2] If absolute and percent inhibition fit in one table results can be unified in one table. |
| | [ ] If absolute and percent initiation in the table results can be unlined in one table. |


200196


Example : Non-Standard \_PD\_T2 Protocol : 2013N167482\_01

Population : PD

Table 3.17
Change from baseline in composite total UAS7 Scores – Comparison

| | | • | |
|---|---|---|---|
| Treatment | N | Mean | Mean Difference vs.<br>Placebo and CI 95% of<br>mean difference |
| Placebo | x | xxx.x | |
| GSK2646264 (0.5%) | X | XXX.X | xx.x (xx.x, xx.x) |
| GSK2646264 (1.0%) | X | XXX.X | xx.x (xx.x, xx.x) |


200196


Example : Non-Standard \_Other\_L1 Protocol : 2013N167482\_01

Population : Safety

Listing 28
Listing of irritation score assessment

| Subject | Treatment | Visit | Irritation<br>Score<br>assessment |
|---------|----------------------|-------|-----------------------------------|
| XXX | GSK2646264<br>(0.5%) | XX | XX |
| | | XX | XX |
| | XXX | XX | XX |

: Non-Standard \_Other\_L2 Page 1 of X : 2013N167482\_01

Protocol : 201 Population : PD

Example

**Listing 31**Listing of Allergen Challenge Parameters

| Treatment | Inv./<br>Subj. | Visit | Parameter<br>(Unit) | Result | Percent o |
|---|---|---|---|---|---|
| XXXXX | XXXXX/<br>XXX | XXXX | XXXXX | XXX.XX | XXX.XX |
| | 7000 | | XXXXX | XXX.XX | XXX.XX |
| | | | XXXXX | XXX.XX | XXX.XX |
| | | | XXXXX | XXX.XX | XXX.XX |
| | | | XXXXX | XXX.XX | XXX.XX |
| | | XXXX | XXXXX | XXX.XX | XXX.XX |
| | | | XXXXX | XXX.XX | XXX.XX |
| | | | XXXXX | XXX.XX | XXX.XX |


Example : Non-Standard \_PD\_F1 Protocol : 2013N167482\_01

Population : PD

Figure 5.1

Allergen Challenge, Weal Area (Percent of Inhibition) - Individual Subject Plot



Programming Notes :

[1] Plot adapted accordingly based on study data (overlayed by treatment)

[2] Subject will have two values one for treatment and another for placebo. Therefore use one colour for the subject id and two symbols for treatment (e.g. o=placebo, +=Treatment). Adapt the graph correspondingly.


Example : Non-Standard \_PD\_F1 Protocol : 2013N167482\_01

Population : PD

Figure 5.2
Allergen Challenge, Weal Area (Percent of Inhibition) - Mean (95% CI) Plot



Treatment: A= Verum, B=Placebo

Programming Notes: [1] Plot adapted accordingly based on study data.
[2] Replicate this box plot to other similar plots, eg. for absolute values..